CLINICAL TRIAL: NCT04102033
Title: Efficacy of Eltrombopag in Chronic Immune Thrombocytopenia in Pediatrics
Brief Title: Eltrombopag in Chronic ITP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, GM Abdelsalam, doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eltrombopag in ITP
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Eltrombopag — Thrombopietic agent approved for its efficacy in chronic immune thrombocytopenia in pediatric patients

SUMMARY:
This study aims to evaluate the efficacy of eltrombopag on the platelet count in pediatric patients with chronic immune thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients with chronic ITP aged 1 to 17 years.
2. Platelet count is less than 30×109 per liter.
3. Patients neither have had spontaneous resolution of the thrombocytopenia nor responded to corticosteroids and/or IV immunoglobulin.

Exclusion Criteria:

1. Patients with clinical and/or laboratory evidence of hepatotoxicity/liver decompensation (Hepatotoxicity due to eltrombopag is defined as increased serum alanine aminotransferase ≥3 times the upper limit of normal (ULN), aspartate aminotransferase ≥3 ULN, alkaline phosphatase >1.5 ULN, total bilirubin >1.5 ULN)
2. Patients with history of thrombotic/thromboembolic events.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Measuring the platelet count response to eltrombopag in pediatric chronic ITP | 6 months

REFERENCES:
- [Background] Corman SL, Mohammad RA. Eltrombopag: a novel oral thrombopoietin receptor agonist. Ann Pharmacother. 2010 Jun;44(6):1072-9. doi: 10.1345/aph.1P042. Epub 2010 May 11. PMID 20460556
- [Background] Bussel JB, de Miguel PG, Despotovic JM, Grainger JD, Sevilla J, Blanchette VS, Krishnamurti L, Connor P, David M, Boayue KB, Matthews DC, Lambert MP, Marcello LM, Iyengar M, Chan GW, Chagin KD, Theodore D, Bailey CK, Bakshi KK. Eltrombopag for the treatment of children with persistent and chronic immune thrombocytopenia (PETIT): a randomised, multicentre, placebo-controlled study. Lancet Haematol. 2015 Aug;2(8):e315-25. doi: 10.1016/S2352-3026(15)00114-3. Epub 2015 Jul 28. PMID 26688484